CLINICAL TRIAL: NCT06798870
Title: Investigation of White Spot Lesions Development During Management of Mixed Dentition Patients with Anterior Functional Shift
Brief Title: White Spot Lesions Development in Mixed Dentition Patients
Acronym: WSL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A0207024OR; A0207024OR (Other: A0207024OR)
Record Dates: First submitted 2024-12-30; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-12

CONDITIONS: Anterior Functional Shift
Keywords: white spot lesion; mixed dentition patients; clear aligner; anterior functional shift
MeSH Terms: interventions — Orthodontic Appliances, Removable

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: blinding the data
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Removable inclined plane group (Active Comparator): removable appliance for correcting anterior crossbite
  Interventions: Device: removable appliances
- clear aligner (Active Comparator): clear aligner appliance for correcting anterior crossbite
  Interventions: Device: removable appliances

INTERVENTIONS:
Device: removable appliances — removable appliances; clear aligner and removable inclined plane, for correcting anterior crossbite vin mixed dentition patient

SUMMARY:
36 patient will be divided into two equal groups. one for removable inclined plane while the other will be treated using clear aligner appliances. evaluation of the white spot lesion will be accumplished for all patients clinically before anr after completion of treatment.

DETAILED DESCRIPTION:
The sample size was calculated using G*Power (Version 3.1.9.4; Germany) and designed to have a power of 82% assuming type I statistical error of 5% and one-tailed statistical test based on Azeem and Hamid.13 The calculated sample was 15 patients in each group. The sample will be increased to include 36 patients: 18 patients per group for a 20% expected loss.

Patients with the age range of 9 to 12 years will be selected for the study. All patients and their parents will be informed of the procedures and will sign the informed consent. Patients who had periodontal diseases, bone resorption cleft lip and palate deformities, orofacial syndrome, hypoplastic enamel defects, and multiple restorations on the facial surfaces or unable to maintain good oral hygiene will be excluded from the study.

All patients will be randomly allocated into two groups according to the management protocol: inclined plane and clear aligner. The patients will be examined for any white spot lesion on the labial surface of the teeth in the upper and lower jaws clinically and using lateral and frontal intraoral photographs immediately before treatment and monthly along the treatment procedures. Each tooth will be evaluated, and the total lesions count will be recorded for each patient. All patients will be instructed to maintain good oral hygiene using fluoridated toothpaste daily.

Statistical analysis:

The incidence of the WSL in each tooth and the total lesions count will be calculated for each patient. These data will be collected and subjected to the appropriate statistical tests using the SPSS version 20.0 software for Windows (IBM, USA).

ELIGIBILITY:
Inclusion Criteria:

* Patients with the age range of 9 to 12 years with anterior crossbite will be selected for the study

Exclusion Criteria:

* periodontal diseases, bone resorption cleft lip and palate deformities, orofacial syndrome, hypoplastic enamel defects, and multiple restorations on the facial surfaces or unable to maintain good oral hygiene

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
development of white spot lesion | 4 months
  examination of the teeth clinically for detecting white spot lesion

SECONDARY OUTCOMES:
the highly incidence of white spot lesion in upper and lower teeth | 4 months
  counting the mostly affected teeth by white spot lesion

CONTACTS AND LOCATIONS:
Overall Officials: NEHAL F Albelasy, PhD, Principal Investigator — Egypt, Mansoura university, faculty of Dentistry, orthodontic department
Locations (1):
- Faculty of Dentistry, Al Mansurah, Egypt